CLINICAL TRIAL: NCT01198223
Title: Comparison of Therapeutic Effect of Aqueous Extract of Garlic and Nystatin Mouthwash in Denture Stomatitis
Brief Title: Effect of Aqueous Extract of Garlic and Nystatin Mouthwash in Denture Stomatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Comparison of therapeutic effect of aqueous extract of garlic and nystatin mouthwash in denture stomatitis, Qazvin University of Medical Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QUMS 1234
Record Dates: First submitted 2010-08-23; First posted 2010-09-10 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-09

CONDITIONS: Denture Stomatitis
Keywords: denture stomatitis; nystatin; garlic
MeSH Terms: conditions — Stomatitis, Denture | interventions — Nystatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- drug: garlic extract, nystatin (Other): Drug: garlic extract 40mg/dl or nystatin suspension 100000 iu/ml tid for one month Patients had been clinically with denture stomatitis and confirmed by oral medicine specialist were selected for the study. Gender, age, medical history, erythema types, size, and other treatment used for this disease were recorded. Local ethical committee approval was obtained before the trial started and all patients gave written informed consent. Patients were randomly divided into two groups .First group received garlic extract and second group used nystatin suspension for 1 month. Each patients was examined at the beginning of the therapy ,and then every 1 weeks up to 1 months .
  Interventions: Drug: garlic , nystatin

INTERVENTIONS:
Drug: garlic , nystatin — mouthwash
  Other Names: aquous garlic

SUMMARY:
The aim of the present study was to compare the effect of aqueous extract of garlic with nystatin mouthwash in denture stomatitis.

DETAILED DESCRIPTION:
Denture stomatitis is the most common form of chronic oral candidiasis manifested as chronic inflammation of the mucous membrane t supporting the movable prosthesis that may have a local or systemic nature. This inflammation is presented as mucous erythema and occasionally with pain and burning. The standard treatment for denture stomatitis is administration of nystatin which is accompanied with complications such as bitter taste as well as the high number of drug application that result in reduced tendency of patients in using this medication hence, efforts are continuously being made to substitute other types of therapies for this condition.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age and older
* confirm of denture stomatitis by the oral medicine specialists

Exclusion Criteria:

* Patients with a history of using anti-fungal drugs, antibiotics, and corticosteroid within the previous month
* allergy to garlic and nystatin mouthwash
* immunodeficiency
* uncontrolled diabetes
* those with garlic rich diet
* inability in using mouthwash
* loose and discolored dentures
* psychologic disorder and alzheimer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
reduction of diameter of erythematous lesion under denture | first week
  measuring erythematous lesion by visual and then photography and a colis

SECONDARY OUTCOMES:
complete relief of erythematous lesions | fourth week

CONTACTS AND LOCATIONS:
Overall Officials: mahin bakhshi, DDS,MS, Study Chair — Qazvin University of Medical Science; Jamileh bigom Taheri, DDS/MS, Study Director — Shahid Beheshti University of Medical Science; Samira Basir Shabestari, DDS/MS, Principal Investigator — QUMS; Rozbeh Pahlevan, DDS, Principal Investigator — QUMS; Anet Tanic, DDS, Principal Investigator — QUMS
Locations (1):
- QUMS, Qazvin, Qazvin Province, Iran